CLINICAL TRIAL: NCT03167437
Title: An Open-Label, Proof of Concept Study of Vorinostat for the Treatment of Moderate-to-Severe Crohn's Disease and Maintenance Therapy With Ustekinumab
Brief Title: An Open-Label, Proof of Consent Study of Vorinostat for the Treatment of Mdoerate-to-Severe Crohn s Disease and Maintenance Therapy With Ustekinumab
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 170101; 17-I-0101
Record Dates: First submitted 2017-05-24; First posted 2017-05-30 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12-23

CONDITIONS: Crohn's Disease
Keywords: Reduce Symptoms of Crohn's Disease; HDAC Inhibitors
MeSH Terms: conditions — Crohn Disease | interventions — Vorinostat; Ustekinumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 1 (Experimental): participants will receive Vorinostat 100mg PO BID for 12 weeks
  Interventions: Drug: Vorinostat
- 2 (Experimental): participants will receive Vorinostat 100mg PO BID for 6months
  Interventions: Drug: Vorinostat
- 3 (Active Comparator): participants will receive ustekinumab (weight base induction dose followed by 90mg SC every 8 weeks for 24 months)
  Interventions: Drug: Ustekinumab

INTERVENTIONS:
Drug: Vorinostat — It is a histone deacetylase (HDAC) inhibitor indicated for the treatment of cutaneous manifestations in patient with cutaneous T-cell lymphoma (CTCL) who have progress, persistent or recurrent disease on or following two systemic therapies. We are using this drug off label for the purpose of this study
  Arms: 1; 2
Drug: Ustekinumab — Ustekinumab inhibits the bioactivity of human IL-12 and IL- 23 by preventing these cytokines from binding to the IL- 12Rbeta1 receptor protein expressed on the surface of immune cells. It is FDA approved for the treatment of adult patients with active psoriatic arthritis and more recently, in September 2016, ustekinumab has been approved for the treatment of patients with Crohn s disease.
  Arms: 3

SUMMARY:
Background:

Crohn s disease (CD) is an inflammatory bowel disease. It causes inflammation of the gut. Symptoms may include diarrhea, abdominal pain, fatigue, weight loss and malnutrition. CD has no cure, but symptoms can sometimes be controlled with medicine. Researchers want to see if it is safe to treat CD with the medicine vorinostat. It is thought that vorinostat may reduce the inflammation process of CD. This may then help to relieve symptoms of CD. Participants who respond to Vorinostat will be invited to an extension phase of treatment with Vorinostat and possibly a maintenance treatment using Ustekinumab.

Objectives:

To see if vorinostat is safe for people with moderate-to-severe CD. To see if it is safe for people with moderate-to-sever CD to receive maintenance therapy using Ustekinumab after successful treatment of Vorinostat.

Eligibility:

Adults 18-65 with moderate-to-severe CD that medicine is not controlling.

Design:

Phase I is screening. It may last 120 days. Participants will have:

Physical exam

Medical history

Tests of blood, urine, and stool samples

Heart test

Questionnaires

Tuberculosis skin test

They may have a colonoscopy and lymphapheresis collection. These will be explained in a separate consent.

They will keep a diary of symptoms.

Phase II is treatment using Vorinostat. It will take 12-13 weeks. Participants will take the study drug by mouth twice daily for 12 weeks. They will get a weekly phone call to talk about how the drug makes them feel. They will have blood taken regularly. Every 4 weeks, they will have a check-up that will repeat some screening tests.

Phase III extension treatment of Vorinostat for an additional 6 months for those who respond to vorinostat and it is safe for them to continue treatment. Participants will continue to receive weekly calls to talk about how the drug makes them feel. They will have blood taken regularly. Every 3 months, they will have a check-up that will repeat some screening tests.

Phase IV: is maintenance therapy for 2 years with Ustekinumab. Participants will receive a one time loading dose of ustekinumab, and then will receive the approved maintenance dose once every 8 weeks, at which time they will return to the NIH Clinical Center for evaluation. The participant will get a phone call 3 days after each dose and again 2 weeks later to see how the drug makes them feel. After two years of receiving treatment with ustekinumab the participant will have an end of study visit, where some of the screening tests, including a colonoscopy, will be repeated.

DETAILED DESCRIPTION:
Crohn s Disease (CD), a major sub-type of inflammatory bowel disease (IBD), is a chronic, life-long condition characterized by relapsing inflammation of the gastrointestinal (GI) tract. Despite recent advances in IBD therapeutics, a significant number of patients with CD continue to have significant symptoms.

In prior studies, it has been demonstrated that epigenetic modifications of the genome are associated with and may contribute to the pathogenesis of various disease entities. One type of epigenetic modification involves acetylation and deacetylation of histones, mediated by histone acetyl transferases (HATs) and histone deacetylases (HDACs). Acetylation and deacetylation of histones regulates the affinity of histones for DNA, thus modulating the accessibility of transcription factors to gene promoters and enhancer sites. Of interest in this context is evidence that epigenetic modifications brought about by HDAC inhibitors (HDACi), i.e., agents that cause hyperacetylation of histones, can limit the course of gastrointestinal inflammation. One naturally occurring HDAC inhibitor, the bacterial product butyrate, has been shown to have effects on gene transcription that regulate potentially deleterious pro-inflammatory responses to microbiota in the gut environment. It has been shown that treatment of dendritic cells and macrophages with butyrate leads to down-regulation of lipopolysaccharide induced pro-inflammatory mediators such as nitric oxide, IL-6 and IL-12. In addition, butyrate has been shown to enhance the differentiation of intestinal Foxp3-positive T cells (T regulatory T cell (Treg) development that then modulates GI inflammation and contributes to mucosal homeostasis. Along the same lines, another HDAC inhibitor, vorinostat, has been shown to ameliorate graft-vs-host disease (GVHD) affecting the GI tract in patients undergoing allogeneic bone marrow transplantation. This anti-inflammatory effect was also attributable to increased Treg activity, suggesting that vorinostat, like butyrate, decreases inflammation by enhancing the activity of cells with the capacity to down- regulate immune responses. The effect of vorinostat on Treg cell expansion in this study was particularly notable because it suggested that Treg cell numbers can be increased by agents that have an intrinsic effect on the transcription of key Treg cell transcription factors. On this basis, treatment of patients with inflammatory and autoimmune diseases by influencing Treg cell numbers may be a more effective than alternative existing methods of inducing Treg cell expansion such as administration of purified Tregs.

In this protocol we propose a proof of concept clinical trial to study the safety and efficacy of vorinostat (100 mg PO BID for 36 weeks) in treating 20 individuals with moderate-to- severe CD who have not been controlled by standard maintenance therapy. This will be accomplished in Phase II (12 weeks of treatment) and Phase III (36 weeks of treatment). We will assess the effectiveness of vorinostat by evaluating changes in symptom scores, endoscopic/histologic findings, and immunologic/laboratory parameters. The participant will return to the NIH CC after starting treatment on week 4, week 8, and week 24 for assessment of safety labs and testing of clinical response. On Week 12 and week 36 participants will return to the NIH CC for assessment of safety labs and testing of clinical and immunologic response.

In Crohn s disease most patients have alternating periods of relapse and remission with half of patients requiring surgery within 10 years of diagnosis on present maintenance therapy. Therefore, the approach to treatment must also evolve from induction control of symptoms to preventing progression of the disease with maintenance therapy. Thus, treatments that safely maintain long-term remission are essential. Treatment guidelines for Crohn s disease recommend maintenance therapy after remission is achieved, particularly for moderate- to-high risk patients. Potential benefits include reduction in hospitalization and surgery and improved quality of life. Long-term efficacy has been studied with azathioprine/mercaptopurine, methotrexate, tumor necrosis factor (TNF) antagonists, and vedolizumab. Although TNF antagonists have significantly advanced the care of Crohn s disease, their efficacy is limited and the development of anti-drug antibodies is associated with loss of response in maintenance therapy. In addition, potential significant side effects of maintenance treatments include bone marrow suppression malignancy and serious infections. Therefore, a need exists for safer agents that have demonstrated improved long-term maintenance efficacy.

The gut inflammation complicating Crohn s disease has been characterized as a T helper type 1 (Th1)/T helper type 17 (Th17) inflammatory response, with excess IL-12, IL-23 cytokine production leading to the generation of excessive IFN-g and IL-17. Ustekinumab, a monoclonal antibody to the p40 subunit of IL-12 and IL-23, is currently FDA approved for the treatment of moderate to severe plaque psoriasis, active psoriatic arthritis, and moderately to severely active CD.

Prior clinical trials have demonstrated long-term efficacy and safety profile of ustekinumab in psoriasis. Similarly, the long-term efficacy and safety of ustekinumab in Crohn s disease dosing had been established in the UNITI trial studies (up to 44 week treatment) in patients who have failed TNF antagonists or other conventional therapies. These studies demonstrated significant response rates and induction of remission rates with a positive safety profile. Studies addressing long term maintenance efficacy of ustekinumab in patients that are in remission have not been performed.

In the present protocol (Phase IV), Crohn s disease patients that have achieved either a defined clinical response or are in remission with vorinostat will then be enrolled to receive long term maintenance treatment with ustekinumab. Participants will receive a weight- based IV loading dose of ustekinumab followed by administration of maintenance doses of 90 mg subcutaneously (SC) every 8 weeks with participants followed over a 2-year period.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Are 18 to 65 years of age, inclusive, at enrollment date.
  2. Have a diagnosis of CD that has been endoscopically or radiographically confirmed. A colonoscopy will be required at baseline to document mucosal disease activity. SES-CD will be obtained with minimum score of 7.
  3. Have active CD symptoms as defined by a CDAI score between 220 and 350 and demonstrate active symptoms as defined by continued weight loss, abdominal pain and/or diarrhea not controlled by standard therapy.
  4. The participant must have active CD symptoms and therefore have had an inadequate response to, loss of response to, or intolerance to at least 1 of the following agent groups in control of their disease (as defined below for each individual agent group: Corticosteroids or Immunomodulators or TNF-alpha sign antagonists or Anti-integrin antibodies)

     a. Corticosteroids

     i. Signs and symptoms of persistently active disease despite a history of at least one 4-week induction regimen that included a dose

     equivalent to prednisone greater than or equal to 30 mg PO once daily (QD) for 2 weeks or intravenously (IV) for 1 week OR

     ii. One failed attempt to taper corticosteroids to below a dose equivalent to prednisone 10 mg PO QD or to taper to below a dose

     of 9 mg of budesonide OR

     iii. History of intolerance of corticosteroids at the discretion of the principal investigator (PI) (including but not limited to Cushing s

     syndrome, osteopenia/osteoporosis, hyperglycemia, insomnia, or infection)

     b. Immunomodulators

     i. Signs and symptoms of persistently active disease despite a history of at least one 12-week regimen of oral azathioprine (AZA) (greater than or equal to 2.5 mg/kg/Day) or 6-MP (greater than or equal to 1.5 mg/kg/Day) OR

     ii. Signs and symptoms of persistently active disease despite a history of at least one 12-week regimen of MTX (greater than or equal to 25 mg/week) OR

     iii. History of intolerance of at least one immunomodulator (including but not limited to nausea/vomiting leading to discontinuation,

     abdominal pain, pancreatitis, liver function test abnormalities, lymphopenia, thiopurine methyltransferase genetic mutation, or

     serious infection)

     c. TNF-alpha sign antagonists with signs and symptoms of persistently active disease despite a history of receiving infliximab, adalimumab, or certolizumab at a dose approved for the treatment of CD and:

     i. Patient had an inadequate response after completing the full induction regimen, per approved product labeling

     ii. Responded initially but then lost response with continued therapy

     iii. Patient had a significant adverse event response which precluded further use including but not exclusion of infusion reaction, serum

     sickness and/or lupus-like rash.

     d. Anti-integrin antibodies: with signs and symptoms of persistently active disease despite a history of receiving an anti-integrin antibody agent (natalizumab or vedolizumab) at a dose approved for the treatment of CD and:

     i. Patient had an inadequate response after completing the full induction regimen, per approved product labeling

     ii. Responded initially but then lost response with continued therapy

     iii. Patient had a significant adverse event response which precluded further use including but not exclusion of infusion reaction, serum

     sickness and/or lupus-like reaction.
  5. At the discretion of the PI, concomitant medications will be permitted if the following conditions are met prior to baseline assessment (Day-1):

     a. 5-aminosalicylic acid (ASA)-based compounds are permissible if:

     i. Oral 5-ASA-based compounds must be at a stable dose for at least 3 weeks prior to baseline or

     ii. Recently discontinued oral 5-ASA-based compounds must have been discontinued at least 3 weeks prior to baseline or

     iii. Rectal 5-ASA-based compounds are not permissible during the study and must have been discontinued at least 3 weeks prior to baseline.

     b. Corticosteroids (e.g., prednisone, budesonide) are permissible if:

     i. Oral corticosteroids must be at a prednisone-equivalent dose of less than or equal to 40 mg/day, or 9 mg/day of budesonide, and have been at a stable dose for at least 3 weeks prior to baseline or

     ii. Discontinuation of oral corticosteroids must have been completed at least 3 weeks prior to baseline or

     iii. Parenteral (subcutaneous, intramuscular, or IV) or rectal corticosteroids are not permitted during the study and must not have been used within a 3-week period prior to baseline

     c. CD-specific antibiotics are permissible if using an antibiotic for treatment of CD ( a CD-specific antibiotic i.e., metronidazole, ciprofloxacin, rifaximin, ampicillin, sulfonamide and tetracycline)

     i. Participants must have been using the antibiotic for at least 3 weeks before baseline at a stable dose or

     ii. If not currently using a CD-specific antibiotic, the stop date must have been at least 3 weeks prior to baseline.

     d. Immunomodulators are permissible if:

     i. Participants receiving chronic (i.e., greater than or equal to 12 weeks) treatment with AZA, 6-MP, or MTX prior to baseline must be on a stable dose for at least 6- 8 weeks prior to baseline and must continue on this same dose during the study. OR

     ii. Participants who have discontinued therapy with AZA, 6-MP, or MTX must have stopped the medication at least 4 weeks prior to baseline. OR

     iii. Participants must not have received therapy with other known immunomodulators (e.g., cyclosporine, tacrolimus, sirolimus, pentoxifylline, or mycophenolate mofetil) or experimental agents (e.g., granulocyte- or macrophage colony stimulating factor) for at least

  8 weeks or 5 half-lives of agent from baseline, whichever is longer.

  e. The use of Anti-TNF and Anti-integrin therapy or other biological therapy listed below will not be permitted and the following washout period will be required in order for participant to be eligible:

  i. Three months washout prior to baseline for certolizumab or natalizumab.

ii. Two months washout prior to baseline for adalimumab, infliximab, and vedolizumab.

iii. 8 week washout prior to baseline for cyclosporine, pimecrolimus, tacrolimus, and any other systemic immunosuppressant.

6. Participants must agree to have samples of their blood and tissue stored for potential future research use.

7. Participants must have a primary medical care provider.

8. Male participants must agree to employ birth control measures to prevent pregnancy in female partners from start of treatment, and continuing through 3 months post treatment.

9. Females of childbearing potential must not be breast-feeding, possibly or actually pregnant, must not have had unprotected intercourse for one month prior to dosing, and must agree not to become pregnant beginning from enrollment in the study to at least 6 months after the end of treatment. Participants must remain completely abstinent of potentially reproductive sexual intercourse (e.g. due to a committed lifestyle) or to consistently use BOTH a barrier method with a spermicide (male or female condom) AND ALSO one of the below listed methods of birth control:

1. Continuous/daily hormonal methods including oral contraceptive pills, patch, implant/injection, etc.
2. Surgical sterilization of either partner, of sufficient duration to be effective, and NOT known to have failed.
3. Intrauterine device.

EXCLUSION CRITERIA:

1. Presence of clinically significant systemic infection (e.g., chronic or acute infection, urinary tract infection, or upper respiratory tract infection) within three months of screening.
2. History or presence of recurrent or chronic infection (e.g., viral infection [including hepatitis B (HBV), hepatitis C (HCV), human immunodeficiency virus (HIV)], bacterial infection, systemic fungal infection, or syphilis).
3. Positive for tuberculosis (TB) via QuantiFERON-Gold (QFT-G). Individuals who are known to have received the tuberculosis vaccine will be administered the QFT- G. Patients can not have received tuberculosis vaccine within 12 months prior to start of study and can not receive tuberculosis vaccine while on study or within 12 months from the time of conclusion of study participation.
4. Has a history of active tuberculosis (TB) or a chest x-ray (CXR) with findings suggestive of old TB infection including calcified nodular lesions, apical fibrosis, or pleural scarring), acute or chronic HBV, HCV, HIV, or opportunistic infections
5. A conduction abnormality on baseline electrocardiogram (ECG) that in the opinion of a cardiologist, is deemed significant.
6. At the discretion of the principal investigator, off-label use of any small molecule therapeutics that are immune modulators (e.g., naltrexone) within 90 days of beginning screening or at any time during the 30 days of the screening window.
7. Presence of abnormal hematological and biochemical parameters, including:

   1. Neutrophil count < 1500 cells/mm3.
   2. Hemoglobin < 9 g/dL.
   3. Platelet count less than or equal to 150,000 cells/mm3.
   4. Creatinine greater than or equal to 1.2 times the upper limit of normal (ULN).
   5. Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) greater than or equal to 1.5 times ULN.
   6. Prothrombin time-international normalized ratio (PT-INR) > 1.0 ULN
   7. Serum bilirubin level > 1.0 times ULN.
8. Individuals on chronic anticoagulation medications.
9. Stool sample positive for GI pathogens potentially causing disease (as assessed by FilmArray GI panel for 22 viral, bacterial, and parasitic organisms that can cause infectious diarrhea [GI pathogen panel]). The principal investigator will consult with an infectious disease specialist to review results and decide whether treatment is warranted.
10. Presence of cytomegalovirus (CMV) infection as defined by positive immunohistochemical staining on tissue intestine biopsy.
11. History of low-grade or high-grade colonic mucosal dysplasia.
12. History of bowel surgery other than perianal (e.g., fistulotomy, seton placement, or abscess drainage) within 6 months prior to beginning the CDAI screening diary or drawing screening blood samples.
13. Presence of surgical changes to gut anatomy that preclude administration of clinical activity indices; this includes but is not limited to ileostomy, colostomy, or subtotal colectomy with ileorectal anastomosis.
14. Known or suspected short bowel syndrome.
15. Requirement of parenteral, total parenteral, elemental oral, or nasogastric nutrition.
16. History or current evidence of cancer, other than non-melanomatous cancer of the skin, or participants that have undergone excision of basal cell carcinoma, squamous cell carcinoma of the skin. All patients receiving ustekinumab will be monitored for the appearance of non-melanoma skin cancer. Patients greater than 60 years of age, those with a medical history of prolonged immunosuppressant therapy and those with a history of PUVA treatment will be followed closely.
17. Unwillingness or inability to comply with study requirements.
18. Presence of only small bowel CD that is inaccessible by standard colonoscopy for harvest of research biopsies. Individuals with only upper gastrointestinal CD or only perianal fistulizing CD are also excluded for this reason.
19. Refusal to abstain from using COX-2 inhibitors or non-steroidal anti-inflammatory drugs (NSAIDs) throughout the study agent administration period.
20. Has uncontrolled diabetes
21. Is taking anti-seizure medication, such as valproic acid or its derivative (i.e., Depakote)
22. Presence of any condition that, in the opinion of the principal investigator, contraindicates participation in this study.
23. Has participated in another investigational trial within 8 weeks (or 5 half-lives of any investigational study agent), whichever is greater, prior to the pre-trial (screening) visit. The window will be derived from the last date of treatment on the previous trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2017-10-30 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of vorinostat in patients with moderate to severe CD as measured by the rate, frequency, and severity of adverse events (AEs) after 12 weeks of treatment. | Days 28, 56 and 12 and 24 weeks after start of treatment
  This is assessing safety issue

SECONDARY OUTCOMES:
170 or greater score on IBDQ | end of Phase III
  Change in Inflammatory Bowel Disease Questionnaire (IBDQ) score from baseline and proportion of participants with a total score of 170 or greater in response to vorinostat.
Determine safety and tolerability of ustekinumab maintenance | end of study
  To determine if ustekinumab is safe and tolerated in CD patients that have received treatment with vorinostat as measured by the rate, frequency, and severity of adverse events (AEs).
Mucosal healing from use of Vorinostat | end of Phase III
  To determine the number of participants with mucosal healing, as assessed by a decrease in endoscopic scores from baseline to zero (Simple Endoscopic Score Crohn s Disease [SES-CD] for CD) or the number of participants with mucosal response as assessed by a decrease from baseline in SES-CD by 50% in response to vorinostat
Changes in CDAI score equal to or greater than 70 | weeks 12 and 24
  To determine the number of participants participants that achievea clinical response at week 12 and week 36, as defined by a decrease in CDAI from baseline by greater than or equal to 70 points for CD patients, upon completion of study Phase II and Phase III
Acheive clinical remission | weeks 12 and 24
  To determine the number of participants that achieve clinical remission at Week 12 and week 36 as defined by a CDAI score of 150 points or less, upon completion of study Phase II and Phase III.
Mucosal healing after ustekinumab maintenance | end of study
  To determine the number of participants with mucosal healing, as assessed by a decrease in endoscopic scores from baseline (vorinostat therapy at week 36) to zero in response to ustekinumab (Simple Endoscopic Score Crohn s Disease [SES-CD] for CD) or the number of participants with mucosal response as assessed by a decrease from baseline in SES-CD by 50% in response to ustekinumab upon completion of Phase IV.
Achieve continued remission with ustekinumab | end of study
  To determine the number of participants that achieve either a continued remission (CDAI < 150) or response after vorinostat therapy at week 36 as defined by a decrease in CDAI from baseline by greater than or equal to 70 points in response to ustekinumab upon completion of Phase IV.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan J Fuss, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Choi SW, Gatza E, Hou G, Sun Y, Whitfield J, Song Y, Oravecz-Wilson K, Tawara I, Dinarello CA, Reddy P. Histone deacetylase inhibition regulates inflammation and enhances Tregs after allogeneic hematopoietic cell transplantation in humans. Blood. 2015 Jan 29;125(5):815-9. doi: 10.1182/blood-2014-10-605238. Epub 2014 Nov 26. PMID 25428224
- [Background] Dinarello CA, Fossati G, Mascagni P. Histone deacetylase inhibitors for treating a spectrum of diseases not related to cancer. Mol Med. 2011 May-Jun;17(5-6):333-52. doi: 10.2119/molmed.2011.00116. Epub 2011 May 5. PMID 21556484
- [Background] Choi SW, Braun T, Chang L, Ferrara JL, Pawarode A, Magenau JM, Hou G, Beumer JH, Levine JE, Goldstein S, Couriel DR, Stockerl-Goldstein K, Krijanovski OI, Kitko C, Yanik GA, Lehmann MH, Tawara I, Sun Y, Paczesny S, Mapara MY, Dinarello CA, DiPersio JF, Reddy P. Vorinostat plus tacrolimus and mycophenolate to prevent graft-versus-host disease after related-donor reduced-intensity conditioning allogeneic haemopoietic stem-cell transplantation: a phase 1/2 trial. Lancet Oncol. 2014 Jan;15(1):87-95. doi: 10.1016/S1470-2045(13)70512-6. Epub 2013 Nov 30. PMID 24295572
- [Derived] Garcia AA, Koperniku A, Ferreira JCB, Mochly-Rosen D. Treatment strategies for glucose-6-phosphate dehydrogenase deficiency: past and future perspectives. Trends Pharmacol Sci. 2021 Oct;42(10):829-844. doi: 10.1016/j.tips.2021.07.002. Epub 2021 Aug 10. PMID 34389161
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2017-I-0101.html